CLINICAL TRIAL: NCT05013775
Title: The Diagnostic Value of Staging Laparoscopy and Computed Tomography Response Assessment in Patients With Gastric Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Sander van Hootegem (Other)
Responsible Party: Sponsor-Investigator, Sander van Hootegem, Investigator, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: MEC-2019-0284
Record Dates: First submitted 2021-08-14; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Tomography, X-Ray Computed; Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Computed tomography — Computed tomography to gauge response after preoperative chemotherapy cycles and excluded the development of interval metastases or irresectable disease
Diagnostic Test: Diagnostic laparoscopy with peritoneal lavage — Diagnostic laparoscopy lavage to exclude (small-volume) metastases and determine local resectability

SUMMARY:
SUMMARY

Rationale: Diagnostic laparoscopy (DL) and response assessment after neoadjuvant chemotherapy with computed tomography (CT) are two diagnostic modalities used to assess metastatic spread in gastric cancer patients. It is still unclear in what proportion of patients clinically relevant metastases or other significant findings (e.g. contra-indications of surgery) are detected that impact on the treatment.

Objective: To determine the clinical value of diagnostic laparoscopy and computed tomography response assessment after neoadjuvant chemotherapy in patients with gastric and esophagogastric junction adenocarcinoma.

Study design: Multicentre retrospective cohort study.

Study population: All Patients with gastric and gastro-oesophageal adenocarcinoma who underwent clinical staging and were discussed at multidisciplinary team meetings (MDT) between January 2016 and December 2018.

Intervention (if applicable): Not applicable.

Main study parameters/endpoints: The main study parameter is the proportion (%) of patients who do not proceed with treatment as planned after a DL and CT response assessment (i.e. the proportion of patients in which metastasized disease or other contra-indications for surgery is found).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Since this is an observational study, no burden or risks are associated with participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven gastric and esophagogastric junction adenocarcinoma.
* Patients who have had (either) DLS and/or CT response assessment (after chemotherapy).
* Discussed at MDT from January 2016 - December 2018
* ≥18 years

Exclusion Criteria:

* Patients with esophagogastric junction adenocarcinoma with the tumour bulk located in the oesophagus that receive neoadjuvant chemoradiation;
* Patients with recurrent/residual disease after earlier treatment of gastric cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with gastric and gastro-oesophageal adenocarcinoma who presented or were referred to one of the participating centres and have been discussed at multidisciplinary team meetings (MDT) for curative management from January 2016 through December 2018. The University Medical Center of the Johannes Gutenberg University Mainz will only contribute with data on DL and not on patients who underwent CT response assessment.
Sampling Method: Non-Probability Sample
Enrollment: 697 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-08-22 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Change in treatment | 1 month (on average)
  Proportion of patients in which the diagnostic test led to change in treatment/management

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided